CLINICAL TRIAL: NCT05753917
Title: Histomorphometric and Immunohistochemical Evaluation of Bone Healing Around Implants Placed Using Piezosurgery Versus Conventional Drills: a Split Mouth Randomized Clinical Trial
Brief Title: Piezo-surgery Versus Conventional Drills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GBR Academy (Network)
Responsible Party: Principal Investigator, Alessandro Cucchi, Alessandro Cucchi, GBR Academy
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16053
Record Dates: First submitted 2023-02-23; First posted 2023-03-03 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Bone Formation
Keywords: piezo-surgery; Implant surgery; histological analysis; Conventional drills

STUDY DESIGN:
Intervention Model Description: Pilot, parallel-group, single-blinded, split-mouth, randomized clinical trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): piezoelectric device with IM1, IM2, IM2-3, or IM3 piezo-inserts according to the manufacturer's protocol (Piezosurgery, Mectron Medical Technology, Carasco, Italy). One or two implants were placed in each edentulous ridge along with an additional 3.3 x 8.5 mm implant, termed a "study fixture", in an adjacent area
  Interventions: Device: Piezo-surgery insert OR Conventional Drills
- Group B (Active Comparator): In Group B, all implant sites were prepared with conventional drills according to the manufacturer's protocol (Premium, Sweden & Martina, Due Carrare, Padova, Italy); similarly to group A, one or two implants were placed in each edentulous ridge, and an additional 3.3 x 8.5 mm "study-fixture" was placed in the adjacent area.
  Interventions: Device: Piezo-surgery insert OR Conventional Drills

INTERVENTIONS:
Device: Piezo-surgery insert OR Conventional Drills — piezo-surgery: Group A (piezoelectric device with IM1, IM2, IM2-3, or IM3 piezo-inserts according to the manufacturer's protocol (Piezosurgery, Mectron Medical Technology, Carasco, Italy) Conventional drill: Group B (conventional drills according to the manufacturer's protocol (Premium, Sweden & Martina, Due Carrare, Padova, Italy)

SUMMARY:
Purpose: The aim of this RCT was to evaluate and compare histomorphometric and immunohistochemical characteristics of peri-implant bone tissue after implant site preparation using piezoelectric tips versus conventional drills. Material and Methods: A split-mouth protocol was carried out on 6 patients with bilateral partial edentulism. A total of 12 alveolar ridges were randomized into two groups: 6 control sites (Group B) with conventional drills preparation (Drill-group) and 6 test sites (Group A) treated by piezoelectric implant inserts preparation (Piezo-group). At 28 days after surgery (T1), in both group, one study-fixtures with 0.5 mm of peri-implant bone tissue were explanted and processed for the histological, histomorphometrical and immunoistochemical analysis. For each sample Inflammatory infiltrates, necrotic bone (Zone 1), woven and newly formed bone (Zone 2), native bone (Zone 3), CD31 (cluster of differentiation 31) and SATB2 (special AT-rich sequence-binding protein necrotic bone undergoing remodeling) were evaluated.

DETAILED DESCRIPTION:
This was a pilot, parallel-group, doble-blinded, split-mouth, randomized clinical trial.

The study included six patients with bilateral partial edentulism, having in total 12 maxillary or mandibular edentulous alveolar ridges. All patients had been referred to the Unit of Oral and Maxillofacial Surgery, Alma Mater Studiorum, University of Bologna, Italy.

The alveolar ridges were randomized into two groups using a computer-generated method: Group A included six regions where implant sites were prepared by piezosurgery, and Group B six regions prepared by conventional drilling.

Surgical and prosthetic protocol In Group A, all implant sites were prepared with a piezoelectric device with IM1, IM2, IM2-3, or IM3 piezo-inserts according to the manufacturer's protocol (Piezosurgery, Mectron Medical Technology, Carasco, Italy). One or two implants were placed in each edentulous ridge along with an additional 3.3 x 8.5 mm implant, termed a "study fixture", in an adjacent area. In Group B, all implant sites were prepared with conventional drills according to the manufacturer's protocol (Premium, Sweden & Martina, Due Carrare, Padova, Italy); similarly to group A, one or two implants were placed in each edentulous ridge, and an additional 3.3 x 8.5 mm "study-fixture" was placed in the adjacent area.

After cover screw placement, a parallel periapical radiograph was taken and the flap was sutured with 4-0 Vicryl. After surgery, antibiotic therapy (1 g amoxicillin and clavulanic acid every 8 h for 4 days), analgesic therapy (nimesulid 200 mg/day for 2 days, continued if pain persisted), and antiseptic therapy (chlorhexidine 0.2% [w/v] three times daily), were prescribed.

* Clinical procedure II - Re-entry Surgery At 28 days after surgery (T1), all "study-fixtures" in both groups were explanted using a trephine drill, taking care to explant the fixture with 0.5 mm of circumferential peri-implant bone tissue. The timing of re-entry surgery (T1) was fixed to be 28 days based on a previous animal study 12. All retrieved implants with bone tissue biopsies were fixed in 4% (v/v) formalin prior to histological analysis (Figure 7,8).
* Clinical procedure III - Prosthetic restoration At 3 months after surgery (T2), a mid-crestal horizontal incisions of keratinized tissue, without vertical incisions, was performed to expose the submerged implants and place healing screws. One month later (T3), implant-supported, metal-ceramic fixed restorations were delivered to the patients to allow functional loading.
* Data collection During surgery and at all postoperative visits (T0, T1, T2, and T3), clinical and radiographic data were recorded by a single operator (E.V.). Histological, histomorphometric, and immunohistochemical data were recorded on the same forms after bone biopsy and laboratory analyses (T1).
* Laboratory data

All specimens were fully analyzed in terms of the percentages of necrotic bone area (NBA%) and newly-formed bone area (nFBA%), and the ratios of these values to total bone area (TBA). For each specimen, the authors identified three different areas proceeding from the surface of the fixture toward the border of the biopsy: zone 1, necrotic bone undergoing remodeling; zone 2, woven and newly formed bone; and zone 3, native bone. For each zone, we recorded:

1. Absolute and relative areas: Zone areas were expressed as absolute values (mm2) and relative values (%) with respect to the total areas.
2. Inflammatory infiltrates: The presence and type of inflammatory infiltrate (if present) was classified; we scored inflammation as absent (no inflammatory cells), minimal (< 5 cells/mm2), or present (> 5 cells/mm2).
3. CD31 (a vascular endothelium differentiation and neo-osteogenesis marker): CD31 expression was recorded as the number of positive vessels/mm2
4. SATB2 (a osteoblastic cell differentiation and osteogenesis marker): SATB2 expression was recorded as the number of positive spots/mm2.

ELIGIBILITY:
Criteria: Inclusion Criteria:

1. bilateral edentulous sites in mandibles or maxillae that did not require bone regeneration prior to implant placement;
2. American Society of Anesthesiologists (ASA) status 1;
3. the capacity to understand and accept the conditions of the study;
4. continuing participation for at least 1 year of follow-up.

Exclusion Criteria:

1. Previous bone augmentation of the sites to be treated;
2. poor oral hygiene;
3. smoking > 10 cigarettes/day;
4. abuse of alcohol or drugs;
5. pregnancy;
6. acute local or systemic infection;
7. uncontrolled diabetes or other metabolic disease;
8. severe hepatic or renal dysfunction;
9. HIV, HBV, or HCV infection;
10. chemotherapy or radiotherapy within the past 5 years;
11. current immunosuppressive therapy;
12. an autoimmune disorder;
13. bisphosphonate therapy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2016-12-12 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2020-12-12 (Actual)

PRIMARY OUTCOMES:
Zone 1 (necrotic bone undergoing remodeling) | after 28 days of healing
  Hystological sections were screened at high magnification (400×), and areas of necrotic bone lacking live osteocytes were automatically outlined with a pointer and photographed using a digital Peltier-cooled camera (Q-color 3; resolution 1,376 x 1,032 pixels; Olympus). Histological and histomorphometric analyses were performed on the central regions of each sample and Image J software (NIH, Bethesda, MD, USA) was used to determine the presence and type of inflammatory infiltrate, and to quantify morphometric parameters. Value expressed as percentage

SECONDARY OUTCOMES:
Zone 2 (woven and newly formed bone) | after 28 days of healing
  Hystological sections were screened at high magnification (400×), and areas of newly formed bone were automatically outlined with a pointer and photographed using a digital Peltier-cooled camera (Q-color 3; resolution 1,376 x 1,032 pixels; Olympus). Histological and histomorphometric analyses were performed on the central regions of each sample and Image J software (NIH, Bethesda, MD, USA) was used to determine the presence and type of inflammatory infiltrate, and to quantify morphometric parameters. Value expressed as percentage
Zone 3 (native bone) | after 28 days of healing
  Hystological sections were screened at high magnification (400×), and areas of native bone were automatically outlined with a pointer and photographed using a digital Peltier-cooled camera (Q-color 3; resolution 1,376 x 1,032 pixels; Olympus). Histological and histomorphometric analyses were performed on the central regions of each sample and Image J software (NIH, Bethesda, MD, USA) was used to determine the presence and type of inflammatory infiltrate, and to quantify morphometric parameters. Value expressed as percentage
CD31 (marker of vascular endothelium differentiation and neo-osteogenesis) | after 28 days of healing
  An automated microscope running "dot slide" software (Olympus Europa SE & Co. KG, Hamburg, Germany) was used to scan all CD31 immunostained slides at 10× magnification to obtain VSI (Virtual Slide Image) files, and the numbers of cells positive for CD31 were counted. CD31 expression was recorded as the number of positive spots/mm2
SATB2 | after 28 days of healing
  An automated microscope running "dot slide" software (Olympus Europa SE & Co. KG, Hamburg, Germany) was used to scan all SATB2 immunostained slides at 10× magnification to obtain VSI (Virtual Slide Image) files, and the numbers of cells positive for SATB2 were counted. SATB2 expression was recorded as the number of positive spots/mm2

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Cucchi, Principal Investigator — GBR Academy

IPD SHARING:
Plan to Share IPD: Yes
Access to the Trial IPD can be requested by qualified researchers engaged in independent scientific research and will be provided following review and approval of a Research Proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA). For more information or to submit a request, please contact dr.cucchi@hotmail.com
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months
Access Criteria: Contact the authors at the following email addresses:
  Alessandro Cucchi: dr.cucchi@hotmail.com Elisabetta Vignudelli: elisabetta.vignudelli@unibo.it